CLINICAL TRIAL: NCT02885116
Title: Hemodynamic Effects of Nasal Highflow on Patients With Chronic Respiratory Insufficiency and Pulmonary Hypertension
Brief Title: Effect of Nasal Highflow on Right Heart Function
Acronym: HÄMOFLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Jens Bräunlich, MD, MD, University of Leipzig
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 461-15-24082015
Record Dates: First submitted 2016-08-22; First posted 2016-08-31 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Pulmonary Hypertension
Keywords: NHF; pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxygen supplementation (Placebo Comparator): right heart catheterization will be done in hypoxemic patients with supplemental oxygen
  Interventions: Device: oxygen supplementation
- Nasal high flow (NHF) supplementation (Active Comparator): right heart catheterization after during NHF (20 min) use with 35 l/min
  Interventions: Device: Nasal high flow (NHF) supplementation

INTERVENTIONS:
Device: Nasal high flow (NHF) supplementation — use of NHF for 20 min/ 35 l/min, at the end of this period right heart catheterization
  Arms: Nasal high flow (NHF) supplementation
Device: oxygen supplementation — hypoxemic patients will use their normal oxygen supplementation durch right heart catheterization
  Arms: oxygen supplementation

SUMMARY:
In this study effect of NHF on pulmonary thermodynamic parameters will studied.

ELIGIBILITY:
Inclusion Criteria:

* stable disease
* hypoxemic respiratory disorder

Exclusion Criteria:

* decompensation
* acute illness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
changes in mean pulmonary pressure (PAPm) | 20 min
  measured in mmHg

SECONDARY OUTCOMES:
changes in wedge pressure (PC) | 20 min
  mmHg
changes in cardiac index (CI) | 20 min
  l/min/qm

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Wirtz, MD, Study Director — Department of Respiratory Medicine
Locations (1):
- Department of Respiratory Medicine, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided